CLINICAL TRIAL: NCT02844140
Title: DE-CT vs. SE-CT as Optimal Imaging During Treatment for Adaptive Proton Therapy in Stage III Non Small Cell Lung Cancer (NSCLC)
Brief Title: DE-CT in Lung Cancer Proton Therapy
Acronym: DE-CT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DE-CT
Record Dates: First submitted 2016-07-19; First posted 2016-07-26 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2016-08

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Scans (Experimental): Patients included in the trial will receive DE-CT in stead of SE-CT's.
  Interventions: Procedure: DE-CT's and SE-CT

INTERVENTIONS:
Procedure: DE-CT's and SE-CT — Patients included in the trial will receive 3 extra DE-CT's and 3 extra SE-CT's

SUMMARY:
Dose distribution calculations for proton therapy are more accurate when based on DE-CT than on SE-CT. It is however unclear what the quantitative benefit of repeated DE-CT calculations is for lung cancer patients.

DETAILED DESCRIPTION:
In order to calculate the dose distribution of protons adequately, accurate estimations of the stopping power ratio (SPR) medium to water, are required. Using a conversion from single energy CT (SE-CT) images results in an uncertainty in the SPR of at least 3-4%. This uncertainty results in in the use of larger margins around the clinical target volume (CTV) and hence more dose to the organs at risk (OAR). It also effects in the conservative use of beam directions, which are often sub-optimal, to avoid irradiating normal tissues.

Dual energy CT (DE-CT) improves the accuracy of the SPR and therefore the proton range estimation.

An evaluation of the proton range for several tissues using SE-CT and DE-CT as input to Monte Carlo (MC) simulations showed on average improvements in range prediction from 0.1% to 2.1% when using DECT instead of SECT, but in several phantoms and also versus proton-CT, the errors on SE-CT based proton stopping power ratios are reported to be more than 7 %.

A limitation of these studies is that most of them were performed in phantoms. In the first clinical data set on five patients with base of skull tumours, it was reported that although the SPR estimation was indeed better for DE-CT than for SE-CT, its clinical relevance was unclear. However, in the same study, phantom measurements showed a large uncertainty of the SPR in the lung. This is due to the large heterogeneity of the lungs and the huge difference in the density of the lungs compared to the mediastinum, the tumour and the chest cavity.

It is therefore important to study the SPR differences of SE-CT compared to DE-CT in lung cancer patients and the impact on the dose distribution especially in the context of adaptive radiotherapy. As during the course of concurrent chemotherapy and radiotherapy, which is the standard treatment in the majority of stage III lung cancer patients, important anatomical changes may occur, it is also of clinical relevance to determine the influence of repeated dose calculations on DE-CT.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced stage IIIA or III B (T0-4 N2-3M0) NSCLC, or M1 oligometastatic disease according to 7th TNM classification.
* Scheduled to receive concurrent chemotherapy and radiotherapy to a dose of at least 60 Gy, as decided at the multidisciplinary tumour board
* Able to give written informed consent
* Able to have adequate contraception in woman with child bearing potential

Exclusion Criteria:

* Not able to give written informed consent
* Not able to comply with adequate contraception in woman with child bearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Dose distribution on the CTV (measured in Gy) | Measured during 2nd and 4th week of radiation treatment
  Dose distribution on the CTV (clinical target volume) of the tumour and the lymph nodes of DE-CT vs. SE-CT
Dose distribution on the OAR (measured in Gy) | Measured during 2nd and 4th week of radiation treatment
  Dose distribution on the OAR (organs at risk), lungs, heart, aorta, pulmonary artery, superior vena cava, oesophagus, spinal cord, vertebral body, of DE-CT vs. SE-CT

CONTACTS AND LOCATIONS:
Overall Officials: Dirk De Ruysscher, MD, PhD, Principal Investigator — Maastro Clinic, The Netherlands
Locations (1):
- MAASTRO clinic, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No